CLINICAL TRIAL: NCT00000367
Title: Prevention of Suicide in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Purpose: Prevention
Other Study IDs: R01MH059366 (NIH); R01MH059366 (NIH); DSIR AT-P
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Depression
Keywords: Depression; Family; Female; Human; Male; Practice Guidelines; Education, Medical, Continuing; Patient Education; Suicide
MeSH Terms: conditions — Depression; Suicide

INTERVENTIONS:
Drug: Treatment of depression
Behavioral: Suicide prevention intervention
Drug: Suicide prevention treatment

SUMMARY:
The purpose of this study is to design a program to prevent suicide in elderly patients by educating patients, their families, and physicians on depression and suicidal thoughts.

A program to prevent suicide in elderly patients needs to be developed. Since elderly patients frequently have doctor's visits, it may be best to have a suicide prevention program based in the patient's doctor's office.

When an older person visits a primary care physician, he/she will check for signs of depression, including thoughts of suicide. The doctor will speak to the patient about depression and how to recognize it. If the individual is diagnosed with depression, the doctor will offer treatment. During this study, the information the doctor collects will be used to evaluate the effectiveness of the program. The study will last for 2 years.

Eligibility for this study is age of at least 60 years and diagnosis of depression. (Depression required for 920 of the 1200 patients; 280 patients should have no symptoms of depression.)

DETAILED DESCRIPTION:
To investigate the effectiveness of an intervention aimed at improving the recognition of suicidal ideation and depression in elderly patients and facilitating the implementation of a treatment algorithm based on the AHCPR (Agency for Health Care Policy and Research) guidelines. To implement procedures aimed at educating patients, families, and physicians on depression and suicidal ideation.

There is a need to test models of depression recognition and treatment to prevent and reduce suicidal behavior in older patients in primary care settings. Elderly suicide most frequently occurs in the context of mild to moderate depression. In primary care patients, suicidal ideation is a risk factor for suicide and has been identified almost exclusively in patients with depressive symptoms and signs. Since most suicide victims are seen by their primary care physicians within a few weeks prior to their death, intervening at the doctor's office may be life-saving.

The intervention is offered in 6 primary care practices from 3 geographic areas (metropolitan and suburban New York, Philadelphia, and Pittsburgh) and its impact is contrasted to that of 6 comparable practices offering usual care. Patients are selected through an age-stratified, two-stage sampling design and followed for 2 years. The group consists of 1,200 subjects and is comprised of patients with depressive symptoms and signs and a random sample of patients without significant depressive symptomatology. Depression Specialists (DS) collaborate with physicians and help them increase recognition, offer timely and appropriately-targeted treatment recommendations, and encourage patients to adhere to treatment. Beyond direct systematic clinical assessment of patients, information is obtained on health services utilization from practice-based medical records and on cause of death from death certificates. Data are also collected to document the impact of intervention on patient care, and on physician knowledge, attitudes, and satisfaction and test hypotheses derived from preliminary studies of the three Intervention Research Centers (IRCs), Cornell, University of Pennsylvania, and University of Pittsburgh, where the study will be conducted.

ELIGIBILITY:
Inclusion Criteria:

-

Patients must have:

Depressive symptoms and signs. (Required for 920 of the 1200 patients; 280 patients should have no significant depressive symptomatology.)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-09; Study Completion 2003-08

CONTACTS AND LOCATIONS:
Overall Officials: George Alexopoulos, MD, Principal Investigator
Locations (1):
- New York Presbyterian Hospital/Westchester Division, White Plains, New York, United States

REFERENCES:
- [Derived] Gallo JJ, Hwang S, Joo JH, Bogner HR, Morales KH, Bruce ML, Reynolds CF 3rd. Multimorbidity, Depression, and Mortality in Primary Care: Randomized Clinical Trial of an Evidence-Based Depression Care Management Program on Mortality Risk. J Gen Intern Med. 2016 Apr;31(4):380-6. doi: 10.1007/s11606-015-3524-y. Epub 2015 Oct 2. PMID 26432693
- [Derived] Gallo JJ, Morales KH, Bogner HR, Raue PJ, Zee J, Bruce ML, Reynolds CF 3rd. Long term effect of depression care management on mortality in older adults: follow-up of cluster randomized clinical trial in primary care. BMJ. 2013 Jun 5;346:f2570. doi: 10.1136/bmj.f2570. PMID 23738992
- [Derived] Gallo JJ, Bogner HR, Morales KH, Post EP, Lin JY, Bruce ML. The effect of a primary care practice-based depression intervention on mortality in older adults: a randomized trial. Ann Intern Med. 2007 May 15;146(10):689-98. doi: 10.7326/0003-4819-146-10-200705150-00002. PMID 17502629